CLINICAL TRIAL: NCT03653767
Title: Effects of Adjustable School Furniture on Health-related Parameters in Students
Brief Title: Effects of Adjustable School Furniture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Primorska (Other)
Collaborators: Innorenew CoE (Other)
Responsible Party: Principal Investigator, Nejc Sarabon, Associate Professor Dr. Sc., University of Primorska
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Classroom Ergonomics
Record Dates: First submitted 2018-08-24; First posted 2018-08-31 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Sedentary Lifestyle
Keywords: classroom ergonomics; sedentary behavior; school interventions; physical activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will use conventional school furniture.
- Adjustable Furniture Group (Experimental): The experimental group will use adjustable ergonomic school furniture.
  Interventions: Device: Adjustable Furniture

INTERVENTIONS:
Device: Adjustable Furniture — The intervention will include adjustable school furniture.
  Arms: Adjustable Furniture Group

SUMMARY:
The aim of this study is to evaluate the level of mismatch between students and school furniture and to assess the effects of adjustable furniture on sedentary behavior, physical activity levels, and sitting posture in students. Firstly, we will obtain the anthropometric measures of all students participating in the study. Secondly, we will calculate the mismatch between the student's anthropometric measures and current school furniture. In the next step, the participants will be separated in two groups, the experimental and the control group. The participants in the experimental group will use adjustable school furniture for one week, whereas the control group will use the conventional school furniture. All the participants will wear an accelerometer for five consecutive days. The results obtained will indicate the furniture mismatch prevalence and demonstrate the effects of adjustable furniture on health-related parameters in students.

DETAILED DESCRIPTION:
Sedentary behavior is a risk factor affecting not only working population but also adolescents. Students spend long period of time seated, which is being associated with reports of musculoskeletal discomfort and pain. The high level of mismatch between students and school furniture is being associated with adolescent lower back pain. The aim of this study is to evaluate the level of mismatch between students and school furniture and to assess the effects of adjustable furniture on sedentary behavior, physical activity levels, and sitting posture in students. Before the experimental part of the study, we will obtain the anthropometric measures of all students participating in the study to calculate the mismatch between the students and the school furniture. In the next step, the participants will be separated to the experimental or the control group. The experimental group will use adjustable school furniture for one week whereas the control group will use the conventional school furniture. All the participants will wear an accelerometer for five consecutive days. The participants will also complete questionnaires about the sedentary behavior and physical activity levels. The sitting posture will be evaluated with Rapid Upper Limb Assessment tool (RULA). Moreover, at the baseline and on the last day of measurements we will measure the classroom environment factors (light, noise, air flow, temperature). The results obtained will indicate the furniture mismatch prevalence and demonstrate the effects of adjustable furniture on health-related parameters in students.

ELIGIBILITY:
Inclusion Criteria:

* aged between 16 and 24 years
* student

Exclusion Criteria:

* body mass index > 30kg/m2
* pain presence in any musculoskeletal part > 3 on 10-level scale
* presence of any non-communicable chronical diseases
* pregnancy

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Change of weekly physical activity levels | 5 days
  Weekly physical activity levels will be measured with accelerometers.
Change of sitting time | 5 days
  Weekly sitting time will be measured with accelerometers.

SECONDARY OUTCOMES:
Adolescent Sedentary Activity Questionnaire | Baseline and after 5 days.
  The Adolescent Sedentary Activity Questionnaire is used to subjectively assess sedentary behavior. Students are asked to think about a normal week, during school term, and to report how long they usually spent engaged in 11 different sedentary behaviors before and after school on each day of the week and on each day of the weekend. If two activities occurred at the same time (e.g., one hour in front of the television doing homework) the students are asked to estimate how much time was spent on each activity during that time (e.g., 45 min television and 15 min homework). Time spent in each category is calculated and time is also summed across categories to yield the total time per week spent in sedentary behavior. Higher outcome values present longer time in sedentary behavior (worse outcome).
Physical Activity Questionnaire for Adolescents | Baseline and after 5 days
  Physical Activity Questionnaire for Adolescents is used to subjectively assess physical activity levels. The questionnaire addresses a habitual week. It consists of three sections, including physical activity in school, during transportation and leisure-time. Each section is further divided into different activity categories. School section: physical education and breaks between lessons. Transportation section: walking and cycling at least 10 minutes at a stretch. Leisure-time section: activities at least 10 min long. A measure of physical activity is then reached by multiplying the time spent for each activity with the corresponding metabolic equivalent (MET-value). Higher outcome value is better, since it indicates a higher level of physical activity and MET values.
Anthropometric measurements of the students performed with anthropometer | Baseline
  Anthropometric measurements will be performed to obtain the main measures that are needed to evaluate the user-furniture mismatch. All the measures will be taken with standard anthropometer, the unit of measure will be centimeter. We will measure Popliteal height, Buttock-popliteal length, Subscapular height, Thigh thickness. Elbow height sitting, Shoulder height sitting. With the measures obtained we will calculate the furniture mismatch for the following: Seat height, Seat depth, Seat to desk clearance, Desk height, Seat width, Upper edge of backrest. Higher percentage of the mismatch between the student's anthropometric measures and furniture indicates a worse outcome.
Sitting posture | Baseline and after 5 days
  The sitting posture will be evaluated with RULA (Rapid Upper Limb Assessment) tool.

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Sarabon, Phd, Principal Investigator — University of Primorska
Locations (1):
- Carpenter High School Skofja Loka, Škofja Loka, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided